CLINICAL TRIAL: NCT00938340
Title: Postprandial Effects of Walnut Components vs Whole Walnuts on Oxidative Stress, Inflammation, Platelet Function, and Endothelial Function in Volunteers With Moderate Hypercholesterolemia
Brief Title: Postprandial Effects of Walnut Components Versus Whole Walnuts on Cardiovascular Disease (CVD) Risk Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PKE 102
Record Dates: First submitted 2009-06-18; First posted 2009-07-13 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Whole walnut (Experimental): 85g whole walnuts, ground, incorporated into inert food carrier
  Interventions: Dietary Supplement: Whole walnut
- Walnut "meat" (Experimental): Separated, ground walnut de-fatted nut meat incorporated into inert food carrier
  Interventions: Dietary Supplement: Walnut "meat"
- Walnut oil (Experimental): Walnut oil extracted from nut meat and incorporated into inert food carrier
  Interventions: Dietary Supplement: Walnut Oil
- Walnut skins (Experimental): Separated, ground walnut skins incorporated into inert food carrier
  Interventions: Dietary Supplement: Walnut Skins

INTERVENTIONS:
Dietary Supplement: Walnut "meat" — Separated, ground walnut de-fatted nut meat incorporated into inert food carrier
  Arms: Walnut "meat"
Dietary Supplement: Walnut Oil — Walnut oil extracted from nut meat and incorporated into inert food carrier
  Arms: Walnut oil
Dietary Supplement: Walnut Skins — Separated, ground walnut skins incorporated into inert food carrier
  Arms: Walnut skins
Dietary Supplement: Whole walnut — 85g whole walnuts, ground, incorporated into inert food carrier
  Arms: Whole walnut

SUMMARY:
The purpose of this study is to evaluate the acute, postprandial effects and mechanism of action of various walnut components (separated nut skins, de-fatted nut meat, nut oil) versus whole walnuts on oxidative stress, inflammation and measures of platelet and endothelial function in healthy adults with moderately elevated cholesterol levels.

DETAILED DESCRIPTION:
Walnuts contain high contents of polyunsaturated fatty acids (PUFA), particularly linoleic acid and linolenic acid. The high PUFA content has been suggested to reduce CVD risk through decreasing total and LDL-cholesterol concentrations, and increasing HDL-C concentrations. In addition, walnuts are rich in substances such as ellagic acid (a polyphenol), antioxidants, vitamin E, fiber, essential fatty acids, flavanoids, and phenolic acids. Polyphenolic compounds are believed to have multiple biological effects influencing oxidative stress, platelet function, inflammation, and cancer initiation and propagation. There is interest in identifying foods with these and other favorable compounds to test their efficacy in real world settings to further understand their role in the human diet. Despite positive benefits found in consumption of the walnuts, it is not known which specific component of the walnut (i.e., whole walnut, walnut skin, defatted walnut, or walnut oil) is most beneficial to health. The investigators hypothesize that maximum improvements in oxidative stress, inflammatory markers, platelet and endothelial function will be observed following consumption of the whole nut versus isolated walnut components, thereby leading to a recommendation to consume walnuts. In addition, results from the research proposed will provide new information about the antioxidant, inflammatory, platelet activity and endothelial effects of the different walnut components and the synergistic effects these components have in the postprandial state.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 60 years
* Body mass index 25-39 kg/m2
* LDL cholesterol >110 mg/dL
* <95 percentile for age and gender for both (based on NHANES data)
* TG < 350 mg/dL

Exclusion Criteria:

* High alcohol consumption > 21 units/week (female subjects) or > 28 units/week (male subjects)
* Intake of vitamin and mineral supplements within the past 3 weeks or unwillingness to discontinue for 3 weeks prior to screening and for entire study.
* Use of prescription cholesterol-lowering or blood pressure-lowering medications during the study
* Intake of other putative cholesterol-lowering supplements (excl. psyllium, fish oil capsules, soy lecithin, phytoestrogens)
* Intake of anti-inflammatory medications (containing aspirin or NSAIDS) on a regular basis or if an acute intake, within 48 hours of a test day
* Diabetes, liver, kidney, thyroid (unless controlled and stable on replacement medication) or other endocrine disorders from self-reported medical history
* Treatment with drugs acting on the gut, such as ezetimibe, bile acid-binding resins, orlistat
* Dietary restrictions such as a medically prescribed diet, or a slimming diet prior to or during the trial
* Weight loss or gain of 10% body weight or more during a period of 6 months before pre-study examination.
* Blood/plasma donation for reason(s) other than the present study prior to the study (1 month for a male subject or 2 months for a female subject), or during the study
* Lactation 6 weeks before the start of and during study, pregnant or wishing to become pregnant 3 months before or during the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State General Clinical Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Berryman CE, Grieger JA, West SG, Chen CY, Blumberg JB, Rothblat GH, Sankaranarayanan S, Kris-Etherton PM. Acute consumption of walnuts and walnut components differentially affect postprandial lipemia, endothelial function, oxidative stress, and cholesterol efflux in humans with mild hypercholesterolemia. J Nutr. 2013 Jun;143(6):788-94. doi: 10.3945/jn.112.170993. Epub 2013 Apr 24. PMID 23616506
- [Derived] Zhang J, Grieger JA, Kris-Etherton PM, Thompson JT, Gillies PJ, Fleming JA, Vanden Heuvel JP. Walnut oil increases cholesterol efflux through inhibition of stearoyl CoA desaturase 1 in THP-1 macrophage-derived foam cells. Nutr Metab (Lond). 2011 Aug 26;8:61. doi: 10.1186/1743-7075-8-61. PMID 21871057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in the local newspaper and university e-mails from April 2008 to October 2008.
Pre-assignment Details: Of the individuals (n=246) who were contacted and screened with a semi-structured telephone interview, 50 qualified and were scheduled for a screening visit at the Penn State General Clinical Research Center. After written informed consent was obtained, a fasting blood sample was drawn. Eligible participants (n=20) were randomized to the study.
Groups:
- Walnut Intervention: Four different treatments were provided to each participant in a randomized-crossover fashion: ground whole walnuts (85 g), walnut skins (5.6 g) derived from whole walnuts, walnut oil (51 g) extracted from whole walnuts, or skinless, defatted walnut nutmeat (34 g) from whole walnuts. Each treatment was incorporated into an inert food carrier.
Period: Overall Study
Arm/Group | Walnut Intervention
Started | 20
Received Whole Walnut Intervention | 16
Received Walnut Nutmeat Intervention | 19
Received Walnut Skins Intervention | 15
Received Walnut Oil Intervention | 15
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Completed Participants (n=15): Whole walnut (85 g) Walnut skins (5.6 g) Walnut oil (51 g) Defatted walnut nutmeat (34 g)
Arm/Group | All Completed Participants (n=15)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29 (4)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 119 (10)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 76 (9)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.0 (0.7)
LDL-cholesterol [Mean (Standard Deviation); unit: mmol/L] | 3.4 (0.6)
HDL-cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.3)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.2 (0.5)
Ferric reducing antioxidant potential (FRAP) [Mean (Standard Deviation); unit: umol TE/L] | 1148 (195)
Total thiols [Mean (Standard Deviation); unit: mmol/L] | 0.40 (0.11)
Malondialdehyde (MDA) [Mean (Standard Deviation); unit: umol/L] | 0.75 (0.32)
Reactive hyperemia index (RHI) [Mean (Standard Deviation); unit: ratio] — RHI was calculated as the ratio of the average pulse wave amplitude during hyperemia (60 to 120 s of the post occlusion period) to the average pulse wave amplitude during baseline in the occluded hand divided by the same values in the control hand and then multiplied by a baseline correction factor.
  ratio | 2.0 (0.6)
Framingham reactive hyperemia index (fRHI) [Mean (Standard Deviation); unit: ln(ratio)] — fRHI is an alternative calculation derived from the same raw data (as RHI) and differs in that it uses the period from 90 to 120 s of postocclusion hyperemia, does not incorporate a baseline correction factor, and has a natural log transformation applied to the resulting ratio.
  ln(ratio) | 0.43 (0.39)

OUTCOME MEASURES:

1. Secondary Outcome: Main Effect of Treatment on Reactive Hyperemia Index (RHI) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. At baseline the endothelial function test was performed using pulse amplitude tonometry (PAT) (Itamar Medical). Participants then had 15 min to consume 1 of the 4 walnut test meals. The endothelial function test was performed again at 240 min postmeal. RHI was calculated as the ratio of the average pulse wave amplitude during hyperemia (60 to 120 s of the post occlusion period) to the average pulse wave amplitude during baseline in the occluded hand divided by the same values in the control hand and then multiplied by a baseline correction factor. No endothelial function test data available for one participant within the walnut oil group and one within the defatted walnut nutmeat group.
Time Frame: Change from baseline at 240 min
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 14 | 14
ratio | -0.19 (0.09) | -0.26 (0.09) | 0.07 (0.09) | -0.09 (0.09)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.012, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g); Test type: Superiority or Other; p = 0.52, Mixed Models Analysis — The Bonferroni adjustment was used to correct for multiple treatment comparisons; P < 0.0083 is considered significant (6 comparisons)
Statistical Analysis 3: Comparison: Whole Walnut (85 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (85 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Walnut Skins (5.6 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Walnut Skins (5.6 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.093, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.12, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

2. Primary Outcome: Main Effect of Treatment on the Ferric Reducing Antioxidant Potential (FRAP) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and FRAP was measured at 0, 60, 120, 240, and 360 min. The FRAP assay was used to determine the reducing ability of plasma in a redox-linked colorimetric reaction. Plasma was incubated with the FRAP reagent at room temperature for 1 h and the absorbance at 593 nm was then recorded. Trolox was used as a reference to construct a standard curve to calculate the FRAP value of the samples. The FRAP assay measures lipophilic and hydrophilic antioxidants (total antioxidant capacity), both of which are present in walnuts.
Time Frame: AUC values were calculated with the trapezoidal rule, using the respective fasting baseline value as the line of reference. Measured at 0 to 360 min (baseline to 360min post meal) for each of the 4 walnut treatments.
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: umol Trolox equivalents (TE)*min/L
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 15 | 15
umol Trolox equivalents (TE)*min/L | -26 (46) | 28 (47) | 9 (47) | -135 (51)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g); Test type: Superiority or Other; p = 0.15, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Whole Walnut (85 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.35, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (85 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Walnut Skins (5.6 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Walnut Skins (5.6 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

3. Primary Outcome: Main Effect of Treatment by Timepoint on the Ferric Reducing Antioxidant Potential (FRAP) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) blood sample was collected. Participants then had 15 min to consume 1 of 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and FRAP was measured at 0, 60, 120, 240, and 360 min. The FRAP assay was used to determine the reducing ability of plasma in a redox-linked colorimetric reaction. Plasma was incubated with the FRAP reagent at room temperature for 1 h and the absorbance at 593 nm was then recorded. Trolox was used as a reference to construct a standard curve to calculate the FRAP value of the samples. The FRAP assay measures lipophilic and hydrophilic antioxidants (total antioxidant capacity), both of which are present in walnuts. Several blood samples (n=3) could not be obtained/measured (walnut skin group at 360 min, walnut oil group at 120 min, whole walnut group at 240 min).
Time Frame: Change from baseline for each timepoint (60, 120, 240, 360 min)
Measure: Least Squares Mean (Standard Error); unit: umol Trolox equivalents (TE)/L
Arm/Group | Whole Walnut (60 Min) | Whole Walnut (120 Min) | Whole Walnut (240 Min) | Whole Walnut (360 Min) | Walnut Skins (60 Min) | Walnut Skins (120 Min) | Walnut Skins (240 Min) | Walnut Skins (360 Min) | Walnut Oil (60 Min) | Walnut Oil (120 Min) | Walnut Oil (240 Min) | Walnut Oil (360 Min) | Defatted Walnut Nutmeat (60 Min) | Defatted Walnut Nutmeat (120 Min) | Defatted Walnut Nutmeat (240 Min) | Defatted Walnut Nutmeat (360 Min)
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15
umol Trolox equivalents (TE)/L | 69 (63) | -34 (63) | -65 (64) | -75 (63) | -4 (64) | 10 (64) | 7 (64) | 98 (65) | -10 (64) | 5 (65) | 53 (64) | -13 (64) | -139 (66) | -92 (66) | -175 (66) | -134 (66)
Statistical Analysis 1: Comparison: Whole Walnut (60 Min) vs Whole Walnut (120 Min) vs Whole Walnut (240 Min) vs Whole Walnut (360 Min) vs Walnut Skins (60 Min) vs Walnut Skins (120 Min) vs Walnut Skins (240 Min) vs Walnut Skins (360 Min) vs Walnut Oil (60 Min) vs Walnut Oil (120 Min) vs Walnut Oil (240 Min) vs Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (60 Min) vs Defatted Walnut Nutmeat (120 Min) vs Defatted Walnut Nutmeat (240 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p = 0.15, Mixed Models Analysis — Main effect of treatment by timepoint

4. Primary Outcome: Main Effect of Treatment on the Changes in Total Thiol Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and total thiols measured at 0, 60, 120, 240, and 360 min. Total thiols in plasma were determined by the following methods: an aliquot of EDTA plasma was mixed with Tris-EDTA buffer, followed by addition of 10 mmol/L 2,2-dithiobisnitrobenzoic acid and methanol. After incubation at room temperature for 15 min and centrifugation, the absorbance of the supernatant was measured at 412 nm.
Time Frame: as for outcome 2
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: mmol*min/L
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmol*min/L | 0.024 (0.014) | 0.010 (0.015) | 0.011 (0.014) | 0.026 (0.017)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.79, Mixed Models Analysis

5. Secondary Outcome: Main Effect of Treatment on Framingham Reactive Hyperemia Index (fRHI) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. At baseline the endothelial function test was performed using pulse amplitude tonometry (PAT) (Itamar Medical). Participants then had 15 min to consume 1 of the 4 walnut test meals. The endothelial function test was performed again at 240 min postmeal. fRHI is an alternative calculation derived from the same raw data (as RHI) and differs in that it uses the period from 90 to 120 s of postocclusion hyperemia, does not incorporate a baseline correction factor, and has a natural log transformation applied to the resulting ratio. No endothelial function test data available for one participant within the walnut oil group and one within the defatted walnut nutmeat group.
Time Frame: Change from baseline at 240 min
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: ln(ratio)
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 14 | 14
ln(ratio) | -0.14 (0.07) | -0.14 (0.07) | 0.09 (0.07) | -0.02 (0.07)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.010, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g); Test type: Superiority or Other; p = 0.98, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Whole Walnut (85 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (85 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Walnut Skins (5.6 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Walnut Skins (5.6 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.16, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Main Effect of Treatment on Heart Rate (HR) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. At baseline the endothelial function test was performed using pulse amplitude tonometry (PAT) (Itamar Medical). Participants then had 15 min to consume 1 of the 4 walnut test meals. The endothelial function test was performed again at 240 min postmeal. No endothelial function test data available for one participant within the walnut oil group and one within the defatted walnut nutmeat group.
Time Frame: Change from baseline at 240 min
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: beats/minute
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 14 | 14
beats/minute | 3.9 (1.4) | 0.2 (1.4) | 4.4 (1.4) | 1.9 (1.5)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.007, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g); Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Whole Walnut (85 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (85 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Walnut Skins (5.6 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Walnut Skins (5.6 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.22, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.074, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

7. Primary Outcome: Main Effect of Treatment by Timepoint on Total Thiol Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and total thiols measured at 0, 60, 120, 240, and 360 min. Total thiols in plasma were determined by the following methods: an aliquot of EDTA plasma was mixed with Tris-EDTA buffer, followed by addition of 10 mmol/L 2,2-dithiobisnitrobenzoic acid and methanol. After incubation at room temperature for 15 min and centrifugation, the absorbance of the supernatant was measured at 412 nm. Several blood samples (n=3) could not be obtained/measured (walnut skin group at 360 min, walnut oil group at 120 min, whole walnut group at 240 min).
Time Frame: Change from baseline for each timepoint (60, 120, 240, 360 min)
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Whole Walnut (60 Min) | Whole Walnut (120 Min) | Whole Walnut (240 Min) | Whole Walnut (360 Min) | Walnut Skins (60 Min) | Walnut Skins (120 Min) | Walnut Skins (240 Min) | Walnut Skins (360 Min) | Walnut Oil (60 Min) | Walnut Oil (120 Min) | Walnut Oil (240 Min) | Walnut Oil (360 Min) | Defatted Walnut Nutmeat (60 Min) | Defatted Walnut Nutmeat (120 Min) | Defatted Walnut Nutmeat (240 Min) | Defatted Walnut Nutmeat (360 Min)
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15
mmol/L | 0.051 (0.017) | 0.035 (0.017) | 0.001 (0.021) | 0.010 (0.022) | 0.018 (0.018) | -0.004 (0.018) | 0.005 (0.021) | 0.019 (0.023) | 0.022 (0.017) | 0.029 (0.018) | 0.003 (0.020) | -0.010 (0.023) | 0.038 (0.019) | 0.037 (0.020) | 0.022 (0.022) | 0.008 (0.024)
Statistical Analysis 1: Comparison: Whole Walnut (60 Min) vs Whole Walnut (120 Min) vs Whole Walnut (240 Min) vs Whole Walnut (360 Min) vs Walnut Skins (60 Min) vs Walnut Skins (120 Min) vs Walnut Skins (240 Min) vs Walnut Skins (360 Min) vs Walnut Oil (60 Min) vs Walnut Oil (120 Min) vs Walnut Oil (240 Min) vs Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (60 Min) vs Defatted Walnut Nutmeat (120 Min) vs Defatted Walnut Nutmeat (240 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p = 0.53, Mixed Models Analysis

8. Primary Outcome: Main Effect of Treatment on the Changes in Malondialdehyde (MDA) Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and MDA measured at 0, 60, 120, 240, and 360 min. Plasma MDA was measured by an Agilent 1100 HPLC system with ﬂuorometric detection.
Time Frame: as for outcome 2
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: umol*min/L
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 15 | 15
umol*min/L | -0.015 (0.036) | 0.004 (0.036) | 0.041 (0.036) | -0.001 (0.037)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

9. Primary Outcome: Main Effect of Treatment by Timepoint on Malondialdehyde (MDA) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the clinic after a 12-h overnight fast. A baseline (0 min) blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and MDA measured at 0, 60, 120, 240, and 360 min. Plasma MDA was measured by an Agilent 1100 HPLC system with ﬂuorometric detection. Several blood samples (n=2) could not be obtained (walnut oil group at 120 min and whole walnut group at 240 min).
Time Frame: Change from baseline for each timepoint (60, 120, 240, 360 min)
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | Whole Walnut (60 Min) | Whole Walnut (120 Min) | Whole Walnut (240 Min) | Whole Walnut (360 Min) | Walnut Skins (60 Min) | Walnut Skins (120 Min) | Walnut Skins (240 Min) | Walnut Skins (360 Min) | Walnut Oil (60 Min) | Walnut Oil (120 Min) | Walnut Oil (240 Min) | Walnut Oil (360 Min) | Defatted Walnut Nutmeat (60 Min) | Defatted Walnut Nutmeat (120 Min) | Defatted Walnut Nutmeat (240 Min) | Defatted Walnut Nutmeat (360 Min)
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15
umol/L | -0.081 (0.056) | -0.018 (0.054) | -0.022 (0.061) | 0.063 (0.075) | -0.054 (0.056) | 0.047 (0.054) | -0.012 (0.060) | 0.049 (0.075) | 0.057 (0.056) | 0.032 (0.056) | -0.021 (0.060) | 0.111 (0.075) | -0.017 (0.056) | 0.004 (0.054) | -0.002 (0.060) | -0.032 (0.075)
Statistical Analysis 1: Comparison: Whole Walnut (60 Min) vs Whole Walnut (120 Min) vs Whole Walnut (240 Min) vs Whole Walnut (360 Min) vs Walnut Skins (60 Min) vs Walnut Skins (120 Min) vs Walnut Skins (240 Min) vs Walnut Skins (360 Min) vs Walnut Oil (60 Min) vs Walnut Oil (120 Min) vs Walnut Oil (240 Min) vs Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (60 Min) vs Defatted Walnut Nutmeat (120 Min) vs Defatted Walnut Nutmeat (240 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

10. Primary Outcome: Main Effect of Treatment on the Changes in C-reactive Protein (CRP) Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and CRP measured at 0, 60, 120, 240, and 360 min. Serum CRP was measured by latex-enhanced immunonephelometry.
Time Frame: as for outcome 2
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: mg*min/L
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 15 | 15
mg*min/L | 0.10 (0.07) | 0.01 (0.07) | 0.20 (0.07) | 0.12 (0.07)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

11. Primary Outcome: Main Effect of Treatment by Timepoint on C-reactive Protein (CRP) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and CRP measured at 0, 60, 120, 240, and 360 min. Serum CRP was measured by latex-enhanced immunonephelometry. Several blood samples (n=3) could not be obtained/measured (walnut oil/120 min, whole walnut/240 min, and walnut skin/360 min).
Time Frame: Change from baseline for each timepoint (60, 120, 240, 360 min)
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Whole Walnut (60 Min) | Whole Walnut (120 Min) | Whole Walnut (240 Min) | Whole Walnut (360 Min) | Walnut Skins (60 Min) | Walnut Skins (120 Min) | Walnut Skins (240 Min) | Walnut Skins (360 Min) | Walnut Oil (60 Min) | Walnut Oil (120 Min) | Walnut Oil (240 Min) | Walnut Oil (360 Min) | Defatted Walnut Nutmeat (60 Min) | Defatted Walnut Nutmeat (120 Min) | Defatted Walnut Nutmeat (240 Min) | Defatted Walnut Nutmeat (360 Min)
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15
mg/L | 0.12 (0.05) | 0.08 (0.05) | 0.06 (0.09) | 0.16 (0.12) | 0.04 (0.06) | 0.03 (0.05) | 0.04 (0.09) | -0.06 (0.13) | 0.20 (0.06) | 0.20 (0.05) | 0.18 (0.09) | 0.25 (0.13) | 0.12 (0.06) | 0.09 (0.06) | 0.08 (0.09) | 0.20 (0.13)
Statistical Analysis 1: Comparison: Whole Walnut (60 Min) vs Whole Walnut (120 Min) vs Whole Walnut (240 Min) vs Whole Walnut (360 Min) vs Walnut Skins (60 Min) vs Walnut Skins (120 Min) vs Walnut Skins (240 Min) vs Walnut Skins (360 Min) vs Walnut Oil (60 Min) vs Walnut Oil (120 Min) vs Walnut Oil (240 Min) vs Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (60 Min) vs Defatted Walnut Nutmeat (120 Min) vs Defatted Walnut Nutmeat (240 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

12. Secondary Outcome: Main Effect of Treatment on Augmentation Index (AI) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. At baseline the endothelial function test was performed using pulse amplitude tonometry (PAT) (Itamar Medical). Participants then had 15 min to consume 1 of the 4 walnut test meals. The endothelial function test was performed again at 240 min postmeal. AI is a measure of vascular stiffness (pulse wave reﬂection) that is calculated from the shape of the pulse wave recorded during baseline. No endothelial function test data was available for one participant within the walnut oil group and one within the defatted walnut nutmeat group.
Time Frame: Change from baseline at 240 min
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 14 | 14
Percent change | -6.6 (3.1) | -1.4 (3.2) | -2.6 (3.2) | -4.0 (3.7)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.44, Mixed Models Analysis

13. Secondary Outcome: Main Effect of Treatment on Augmentation Index Standardized to a Heart Rate of 75 Beats/Min (AI_75) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. At baseline the endothelial function test was performed using pulse amplitude tonometry (PAT) (Itamar Medical). Participants then had 15 min to consume 1 of the 4 walnut test meals. The endothelial function test was performed again at 240 min postmeal. AI is a measure of vascular stiffness (pulse wave reﬂection) that is calculated from the shape of the pulse wave recorded during baseline. AI can be adjusted to a heart rate of 75 beats/min (AI_75) to correct for the independent effect of heart rate on this measure.No endothelial function test data was available for one participant within the walnut oil group and one within the defatted walnut nutmeat group.
Time Frame: Change from baseline at 240 min
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 14 | 14
Percent change | -4.0 (2.7) | -1.2 (2.8) | -0.1 (2.9) | -2.9 (3.3)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis

14. Secondary Outcome: Main Effect of Treatment on the Triglyceride (TG) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and TG was measured at 0, 30, 60, 120, 240, and 360 min. TG were determined by standard colorimetric and enzymatic procedures with commercially available kits (Alfa Wassermann).
Time Frame: as for outcome 2
Population: All participants who completed each of the 4 treatment arms
Measure: Least Squares Mean (Standard Error); unit: mmol*min/L
Arm/Group | Whole Walnut (85 g) | Walnut Skins (5.6 g) | Walnut Oil (51 g) | Defatted Walnut Nutmeat (34 g)
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmol*min/L | 0.24 (0.05) | 0.05 (0.05) | 0.24 (0.05) | 0.09 (0.06)
Statistical Analysis 1: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g) vs Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.011, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (85 g) vs Walnut Skins (5.6 g); Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Whole Walnut (85 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (85 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.037, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Walnut Skins (5.6 g) vs Walnut Oil (51 g); Test type: Superiority or Other; p = 0.0087, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Walnut Skins (5.6 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.64, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Walnut Oil (51 g) vs Defatted Walnut Nutmeat (34 g); Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

15. Secondary Outcome: Main Effect of Treatment by Timepoint on Triglyceride (TG) Changes in Response to 4 Walnut Treatments
Description: On the day of each test, participants arrived at the General Clinical Research Center after a 12-h overnight fast. A baseline (0 min) fasting blood sample was collected. Participants then had 15 min to consume 1 of the 4 walnut test meals. Blood samples (∼30 mL) were subsequently taken at 30, 60, 120, 240, and 360 min following the meal and TG was measured at 0, 30, 60, 120, 240, and 360 min. TG were determined by standard colorimetric and enzymatic procedures with commercially available kits (Alfa Wassermann). Several blood samples (n=4) could not be obtained/measured [walnut skin group at 360 min (n=1), walnut oil group at 120 min (n=2), whole walnut group at 240 min(n=1)].
Time Frame: Change from baseline for each timepoint (30, 60, 120, 240, 360 min)
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Whole Walnut (30 Min) | Whole Walnut (60 Min) | Whole Walnut (120 Min) | Whole Walnut (240 Min) | Whole Walnut (360 Min) | Walnut Skins (30 Min) | Walnut Skins (60 Min) | Walnut Skins (120 Min) | Walnut Skins (240 Min) | Walnut Skins (360 Min) | Walnut Oil (30 Min) | Walnut Oil (60 Min) | Walnut Oil (120 Min) | Walnut Oil (240 Min) | Walnut Oil (360 Min) | Defatted Walnut Nutmeat (30 Min) | Defatted Walnut Nutmeat (60 Min) | Defatted Walnut Nutmeat (120 Min) | Defatted Walnut Nutmeat (240 Min) | Defatted Walnut Nutmeat (360 Min)
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 14 | 15
mmol/L | 0.04 (0.04) | 0.13 (0.05) | 0.32 (0.07) | 0.47 (0.08) | 0.24 (0.07) | 0.05 (0.04) | 0.05 (0.05) | 0.02 (0.07) | 0.06 (0.08) | 0.08 (0.07) | 0.08 (0.04) | 0.10 (0.05) | 0.41 (0.07) | 0.47 (0.08) | 0.14 (0.07) | 0.05 (0.05) | 0.02 (0.06) | 0.06 (0.07) | 0.17 (0.09) | 0.13 (0.08)
Statistical Analysis 1: Comparison: Whole Walnut (30 Min) vs Whole Walnut (60 Min) vs Whole Walnut (120 Min) vs Whole Walnut (240 Min) vs Whole Walnut (360 Min) vs Walnut Skins (30 Min) vs Walnut Skins (60 Min) vs Walnut Skins (120 Min) vs Walnut Skins (240 Min) vs Walnut Skins (360 Min) vs Walnut Oil (30 Min) vs Walnut Oil (60 Min) vs Walnut Oil (120 Min) vs Walnut Oil (240 Min) vs Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (30 Min) vs Defatted Walnut Nutmeat (60 Min) vs Defatted Walnut Nutmeat (120 Min) vs Defatted Walnut Nutmeat (240 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Whole Walnut (30 Min) vs Walnut Skins (30 Min); Test type: Superiority or Other; p = 0.91, Mixed Models Analysis — The Bonferroni adjustment was used to correct for multiple treatment comparisons; P < 0.001667 is considered significant (30 comparisons)
Statistical Analysis 3: Comparison: Whole Walnut (60 Min) vs Walnut Skins (60 Min); Test type: Superiority or Other; p = 0.21, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 4: Comparison: Whole Walnut (120 Min) vs Walnut Skins (120 Min); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 5: Comparison: Whole Walnut (240 Min) vs Walnut Skins (240 Min); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 6: Comparison: Whole Walnut (360 Min) vs Walnut Skins (360 Min); Test type: Superiority or Other; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 7: Comparison: Whole Walnut (30 Min) vs Walnut Oil (30 Min); Test type: Superiority or Other; p = 0.53, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 8: Comparison: Whole Walnut (60 Min) vs Walnut Oil (60 Min); Test type: Superiority or Other; p = 0.59, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 9: Comparison: Whole Walnut (120 Min) vs Walnut Oil (120 Min); Test type: Superiority or Other; p = 0.31, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 10: Comparison: Whole Walnut (240 Min) vs Walnut Oil (240 Min); Test type: Superiority or Other; p = 0.98, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 11: Comparison: Whole Walnut (360 Min) vs Walnut Oil (360 Min); Test type: Superiority or Other; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 12: Comparison: Whole Walnut (30 Min) vs Defatted Walnut Nutmeat (30 Min); Test type: Superiority or Other; p = 0.91, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 13: Comparison: Whole Walnut (60 Min) vs Defatted Walnut Nutmeat (60 Min); Test type: Superiority or Other; p = 0.12, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 14: Comparison: Whole Walnut (120 Min) vs Defatted Walnut Nutmeat (120 Min); Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 15: Comparison: Whole Walnut (240 Min) vs Defatted Walnut Nutmeat (240 Min); Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 16: Comparison: Whole Walnut (360 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p = 0.28, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 17: Comparison: Walnut Skins (30 Min) vs Walnut Oil (30 Min); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 18: Comparison: Walnut Skins (60 Min) vs Walnut Oil (60 Min); Test type: Superiority or Other; p = 0.48, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 19: Comparison: Walnut Skins (120 Min) vs Walnut Oil (120 Min); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 20: Comparison: Walnut Skins (240 Min) vs Walnut Oil (240 Min); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 21: Comparison: Walnut Skins (360 Min) vs Walnut Oil (360 Min); Test type: Superiority or Other; p = 0.57, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 22: Comparison: Walnut Skins (30 Min) vs Defatted Walnut Nutmeat (30 Min); Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 23: Comparison: Walnut Skins (60 Min) vs Defatted Walnut Nutmeat (60 Min); Test type: Superiority or Other; p = 0.71, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 24: Comparison: Walnut Skins (120 Min) vs Defatted Walnut Nutmeat (120 Min); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 25: Comparison: Walnut Skins (240 Min) vs Defatted Walnut Nutmeat (240 Min); Test type: Superiority or Other; p = 0.33, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 26: Comparison: Walnut Skins (360 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p = 0.65, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 27: Comparison: Walnut Oil (30 Min) vs Defatted Walnut Nutmeat (30 Min); Test type: Superiority or Other; p = 0.66, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 28: Comparison: Walnut Oil (60 Min) vs Defatted Walnut Nutmeat (60 Min); Test type: Superiority or Other; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 29: Comparison: Walnut Oil (120 Min) vs Defatted Walnut Nutmeat (120 Min); Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 30: Comparison: Walnut Oil (240 Min) vs Defatted Walnut Nutmeat (240 Min); Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]
Statistical Analysis 31: Comparison: Walnut Oil (360 Min) vs Defatted Walnut Nutmeat (360 Min); Test type: Superiority or Other; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]

ADVERSE EVENTS:
Time Frame: During the intervention (0 to 360 min)
Arm/Group | Walnut Oil | Whole Walnut | Walnut Skins | Defatted Walnut Nutmeat
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 0/15 | 0/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walnut Oil (N=15) | Whole Walnut (N=15) | Walnut Skins (N=15) | Defatted Walnut Nutmeat (N=15)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No